CLINICAL TRIAL: NCT04230135
Title: Randomised Controlled Trial to Test to What Extent the Adaptation of a Smartphone-based Self-help Programme to Albanian Immigrants' Cultural Concepts of Distress Enhances Its Acceptability and Efficacy
Brief Title: Cultural Adaptation of Hap-pas-Hapi (Step-by-Step) for Albanian-speaking Immigrants in Switzerland and Germany
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An insufficient number of participants could be recruited, and drop-out rates were very high (80%)
Sponsor: University of Zurich (Other)
Collaborators: Freie Universität Berlin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hap-pas-Hapi
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Psychological Distress

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generic (surface adaptation) (Active Comparator): The generic version of Hap-pas-Hapi includes only surface adaptations (i.e., adaptation of text and illustrations that are inacceptable or non-meaningful for the target group)
  Interventions: Device: Hap-pas-Hapi
- Adapted (deep structure adaptation) (Experimental): For the experimental intervention, Hap-pas-Hapi was adapted to Albanian immigrants' cultural concepts of distress (CCD). An ethnopsychological study was conducted for this purpose, since evidence on CCD in South Eastern Europe is scarce. Based on this study, three deep-structure adaptations were done: i) the symptom narrative provided by the narrator in the app was re-written to reflect Albanian immigrants' CCD; ii) a new explanatory model builder was implemented to address the target group's fatalistic beliefs; and iii) a goal-setting task was programmed to address the target group's socio-centric notion of the self.
  Interventions: Device: Hap-pas-Hapi

INTERVENTIONS:
Device: Hap-pas-Hapi — Hap-pas-Hapi is a Smartphone-based intervention for the treatment of psychological distress. It includes five sessions and uses a narrative approach. Behavioural activation is the main active therapeutic agent in the intervention, along with stress management, positive self-talk, mood tracking, social support, and relapse prevention.

SUMMARY:
We aim to compare two different levels of cultural adaptation of an Internet- and mobile-based intervention for the treatment of depression called Hap-pas-Hapi among Albanian-speaking immigrants in Switzerland and Germany. One arm will include the generic (minimally adapted) version of Hap-pas Hapi. The other arm will include a version of Hap-pas-Hapi that was adapted to the target population's cultural concepts of distress. Both versions include five sessions and the same therapeutic techniques.

ELIGIBILITY:
Inclusion Criteria:

* Electronic informed consent documented by time-stamped agreement to a set of consent questions
* Albanian-speaking
* Male and female participants aged above 18
* Kessler Psychological Distress Scale (K10), Albanian version score >15
* Access to Smartphone (iOS or Android) or web-browser

Exclusion Criteria:

* People living outside Germany or Switzerland
* Serious suicidal thoughts or plan (self-assessed with a corresponding question)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Psychological distress | Six weeks
  Hopkins Symptom Checklist-25 (HSCL-25)
Treatment adherence | Six weeks
  Completing at least three (out of five) sessions of Hap-pas-Hapi;

SECONDARY OUTCOMES:
Functional impairment (health and disability) | Six weeks
  WHO Disability Assessment Schedule (WHODAS 2.0)
Well-being | Six weeks
  The WHO Wellbeing Index (WHO-5)
Post-traumatic stress disorder | Six weeks
  The PTSD checklist, 8 items version (PCL-8)
Self-defined problems | Six weeks
  The Psychological Outcome Profiles (PSYCHLOPS)

CONTACTS AND LOCATIONS:
Locations (2):
- Freie Universität Berlin, Berlin, Germany
- University of Zurich, Zurich, Switzerland